CLINICAL TRIAL: NCT05349825
Title: Investigation of MDR1 (Multi-Drug Resistance) Gene Polymorphism and Losartan Plasma Concentration in Patients Undergoing Hypertensive Episodes While Under Losartan Treatment: A Prospective, Case-Control Study
Brief Title: Investigation of MDR1 Gene Polymorphism and Losartan Plasma Concentration in Patients Undergoing Hypertensive Episodes While Under Losartan Treatment
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Üzeyir Çimen, Research Assistant, Pamukkale University
Other Study IDs: 4921
Record Dates: First submitted 2022-04-18; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Hypertension
Keywords: Losartan; MDR1; Genetic polymorphism; EXP3174; Hypertension
MeSH Terms: conditions — Hypertension | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — 20 ml of blood was collected from the enrolled patients. 10 ml of blood was stored in the tubes with ethylene diamine tetraacetic acid (EDTA) until Deoxyribonucleic acid (DNA) isolation was performed at -20 degrees and plasma level was identified. The remaining 10 ml was centrifuged at 3500 rpm for 10 min, and the plasma was separated. The resulting plasmas were stored in the eppendorf tubes at -20°C until the tandem mass spectrometry measurement
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Hypertensive episode: 50 individuals presenting with a hypertensive episode (patients under 60, >140/90 mmHg, patients over 60, >150/90 mmHg, according to the JNC8 guidelines) while under losartan treatment
  Interventions: Diagnostic Test: Genetic analysis and Losartan plazma level measurement
- Patients with controlled hypertension: 50 patients whose blood pressure was regulated while receiving losartan treatment and who were admitted to the ED for reasons other than hypertensive episode. The eligible patients matching the inclusion and exclusion criteria were recruited for the study.
  Interventions: Diagnostic Test: Genetic analysis and Losartan plazma level measurement

INTERVENTIONS:
Diagnostic Test: Genetic analysis and Losartan plazma level measurement — 20 ml of blood was collected from the enrolled patients. 10 ml of blood was stored in the tubes with ethylene diamine tetraacetic acid (EDTA) until Deoxyribonucleic acid (DNA) isolation was performed at -20 degrees and plasma level was identified. The remaining 10 ml was centrifuged at 3500 rpm for 10 min, and the plasma was separated. The resulting plasmas were stored in the eppendorf tubes at -20°C until the tandem mass spectrometry measurement. The blood samples in EDTA tubes were then transferred for DNA analysis. . To measure plasma losartan concentration, after the frozen plasma samples stored in the eppendorfs were thawed and brought to room temperature, plasma losartan and EXP3174 levels of the patients were calculated using tandem mass spectrometry

SUMMARY:
Losartan is an antihypertensive drug belonging to the ARB family. It is characterized as the substrate of the Multi Drug Resistance-1 (MDR1) drug-efflux protein (a pump that ensures the removal of drugs/foreign substances out of the cell) encoded by the ATP Binding Cassette Subfamily B Member 1 (ABCB1) gene. A recent line of evidence indicates that potential polymorphisms in this gene tend to alter the absorption, transport, bioavailability of losartan, and, indirectly, its effectiveness in hypertension control. As identified by new research, the C3435T, G2677T, and C1236T polymorphic alleles of the MDR1 gene might alter the bioavailability and thus the effectiveness of losartan

DETAILED DESCRIPTION:
This trial was conducted in the emergency services of Gazi University and Pamukkale University. The patient group was comprised of 50 individuals presenting with a hypertensive episode (patients under 60, >140/90 mmHg, patients over 60, >150/90 mmHg, according to the JNC8 guidelines) while under losartan treatment. The control group, by contrast, included 50 patients whose blood pressure was regulated while receiving losartan treatment and who were admitted to the ED for reasons other than hypertensive episode. The eligible patients matching the inclusion and exclusion criteria were recruited for the study.

Within the scope of this research, we included hypertension patients over 18 who gave their informed consent for the study and received minimum 25 mg losartan daily for at least six weeks. 50 individuals admitted to the ED due to a hypertensive episode while under losartan treatment were assigned to the patient group, while 50 patients whose blood pressure was regulated while receiving losartan treatment and who were admitted to the ED for reasons other than hypertensive episode were included in the control group. Those who did not give their consent to participate and did not match the inclusion criteria were excluded from the scope of the study Prior to the trial, the participants were assessed based on the pre-defined patient selection criteria, and the non-eligible ones were excluded from the trial. These exclusion criteria can be listed as refusal to participate in the study, illiteracy, being under 18, being pregnant and in lactation period, being hemodynamically unstable (mean arterial pressure <65mmHg), undergoing kidney transplantation, having liver failure (CHILD PUGH Class C and higher patients) or renal failure (GFR<60), and taking anti-hypertensive drugs other than losartan(Figure 1).

Initially, 20 ml of blood was collected from the enrolled patients. 10 ml of blood was stored in the tubes with ethylene diamine tetraacetic acid (EDTA) until Deoxyribonucleic acid (DNA) isolation was performed at -20 degrees and plasma level was identified. The remaining 10 ml was centrifuged at 3500 rpm for 10 min, and the plasma was separated. The resulting plasmas were stored in the eppendorf tubes at -20°C until the tandem mass spectrometry measurement.

ELIGIBILITY:
Inclusion Criteria:

* gave their informed consent
* received minimum 25 mg losartan daily for at least six weeks

Exclusion Criteria:

* refusal to participate in the study
* illiteracy
* pregnant or in lactation period
* hemodynamically unstable (mean arterial pressure <65mmHg)
* kidney transplantation
* liver failure (CHILD PUGH Class C and higher patients) or renal failure (GFR<60)
* taking anti-hypertensive drugs other than losartan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: . The patient group was comprised of 50 individuals presenting with a hypertensive episode (patients under 60, >140/90 mmHg, patients over 60, >150/90 mmHg, according to the JNC8 guidelines) while under losartan treatment. The control group, by contrast, included 50 patients whose blood pressure was regulated while receiving losartan treatment and who were admitted to the ED for reasons other than hypertensive episode.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
MDR1 gene polimorphism does not influence losartan consantration nevertheless changes blood pressure lowering effect of losartan | at least six weeks under losartan treatment
  50 patients receiving anti-hypertensive treatment with losartan, presenting to the ED with a hypertensive episode and 50 patients whose blood pressure was regulated while receiving losartan treatment and who presented to the ED for reasons other than hypertensive episode. Compare two groups losartan consantration and MDR1 gene polymorphyms

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided